CLINICAL TRIAL: NCT07368985
Title: A Phase II Single Arm Open Label Study of Pembrolizumab and Lenvatinib in Patients With High Risk Locally Advanced Cervix Cancer: an EMBRACE High Risk Study Initiative
Brief Title: Pembrolizumab and Lenvatinib in Patients With High Risk Locally Advanced Cervix Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dr. Remi A. Nout (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Prof. Dr. Remi A. Nout, Professor, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-506982-73-00; 2023-506982-73-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-22; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Cervical Cancer by FIGO Stage 2018; Squamous Cell Carcinoma FIGO 2018 Stage IIIA, IIIB, IIIC1-IIIC2; Adenocarcinoma or Adeno-squamous Carcinoma Stage IB3-IIIC2
Keywords: cervical cancer; locally advanced cervical cancer; Pembrolizumab; Lenvatinib; radiotherapy; brachytherapy; high risk locally advanced cervical cancer
MeSH Terms: conditions — Adenocarcinoma; Uterine Cervical Neoplasms | interventions — pembrolizumab; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Single arm: Pembrolizumab and Lenvatinib (Experimental): Single arm open label study of Pembrolizumab and Lenvatinib in patients with high risk locally advanced cervix cancer that will undergo chemoradiation and brachytherapy
  Interventions: Drug: pembrolizumab and lenvatinib

INTERVENTIONS:
Drug: pembrolizumab and lenvatinib — Patients will undergo standard of care chemoradiation (CRT: combined external beam radiotherapy with weekly cisplatin) followed by MRI guided brachytherapy, this will be combined with the following study drugs:
  Pembrolizumab: 5 intravenous administrations of Pembrolizumab (200 mg) every 3 weeks with the first administration at the start of chemoradiotherapy, followed by subsequent doses of 400 mg IV Pembrolizumab at 6 weeks intervals, starting week 16 up to week 102 with a maximum of 15 cycles.
  Lenvatinib: the combination with Lenvatinib will start after recovery, along with the 6 weekly cycles of Pembrolizumab, e.g. around 8-9 weeks after brachytherapy (week 16), at a dose of 20 mg daily oral and will continue up to week 48.

SUMMARY:
The goal of this clinical trial is to learn if the combination of Pembrolizumab and Lenvatinib works to treat locally advanced cervical cancer in adults that will undergo primary chemoradiation and brachytherapy. It will also learn about the safety of the combination of Pembrolizumab and Lenvatinib. The main questions it aims to answer are:

* Does the combination of Pembrolizumab and Lenvatinib improve progression free survival at two years after treatment?
* What side effects do participants have when taking the combination of Pembrolizumab and Lenvatinib? Researchers will compare the combination of Pembrolizumab and Lenvatinib to existing results with primary chemoradiatoin and brachytherapy to see if the combination of Pembrolizumab and Lenvatinib works to treat locally advanced cervical cancer.

Participants will:

* Visit the clinic to receive Pembrolizumab intra venously once every 3 weeks for 5 cycles and then once very 6 weeks for a maximum of 2-years
* Take Lenvatinib orally every day starting at the earliest 8 weeks after the last brachytherapy to a maximum of 1 year
* Visit the clinic for checkups and tests during scheduled visits

DETAILED DESCRIPTION:
Rationale Chemoradiation (CRT: combined external beam radiotherapy with weekly cisplatin) followed by brachytherapy has remained the standard first line treatment for locally advanced cervical (LACC) patients. Over the last decades, major improvements in radiotherapy have been pioneered through the EMBRACE studies. Most recently the outcome data of 1318 patients undergoing response adapted advanced MRI image guided intracavitary +/-interstitial brachytherapy (MR-IGABT) over and above CRT have been reported. This dose escalated approach resulted in 5-year local control of 92%, pelvic control of 87% and disease-free survival (DFS) of 68%. In this cohort, a 5-year OS of 64% was observed for stage IIIB and 67% for node positive patients. These results essentially confirm both the effectiveness of MR-IGABT for pelvic control but also the need of more effective systemic therapy approaches. Patients most at risk for recurrence and reduced 3-year DFS include patients with presence of multiple nodes in pelvic and paraaortic region or adeno/adenosquamous carcinoma histological type and those with a poor response to CRT.

Considering that both anti-angiogenesis and immune checkpoint blockade work independently in cervix cancer, a combination approach may be associated with synergy and improved outcomes. Recently, the phase III randomized placebo-controlled KEYNOTE A-18 trial investigated the combination of CRT with anti-PD-1 Pembrolizumab in patients with high-risk locally advanced cervical cancer defined as FIGO 2014 stage IB2-IIB with node-positive disease or stage III-IVA regardless of nodal status. With a median follow-up of 17·9 months a 11% progression free survival (PFS) benefit at 2-years was demonstrated (68% vs 57%). Timing immunotherapy during radiotherapy and close to brachytherapy (where high dose per fraction is utilised) may allow to maximally synchronize "immunotherapy response" by taking advantage of the "inflamed" tumour microenvironment and a high radiotherapy dose fraction that is administered using brachytherapy. Lenvatinib will be initiated not earlier than 8 weeks after the last CRT and brachytherapy, to allow for sufficient healing of acute side effects of CRT.

The study hypothesizes that over and above concurrent and Pembrolizumab monotherapy, the addition of Lenvatinib administered after CRT and brachytherapy will lead to improved outcomes in this high-risk population of patients with locally advanced cervical cancer.

Objective The primary objective of the trial is to evaluate progression free survival (PFS) at 24 months (by investigator assessed RECIST 1.1) in women with high-risk locally advanced cervical cancer treated with chemoradiotherapy and Pembrolizumab followed by Pembrolizumab and Lenvatinib. Secondary Objectives include overall survival (OS), local and regional control; physician reported toxicity (CTCAE v5.0) and patient reported outcomes (EORTC QLQ-C30 and CX-24); and associated tissue, blood and imaging based translational research.

Interventions Patients will undergo standard of care chemoradiation (CRT: combined external beam radiotherapy with weekly cisplatin). Initial tumor imaging at pre-screening must have been performed within 28 days prior to the date of registration. The site study team must review pre-treatment images to confirm the participant has measurable disease per RECIST 1.1 at diagnosis. Target definition and dose reporting follow ICRU-89 and are detailed in the protocol. The elective node target volume is risk based and follows EMBRACE-II, that includes elective para-aortic radiotherapy up to the crossing of the renal vessels in patients with: ≥ 1 pathologic node at common iliac or above OR ≥ 3 pathologic nodes. With regard to organs at risk (OAR) for bowel the outer loops are contoured including the mesenteric, and for bones the whole bone from ischial tuberosity to 25mm superior of the PTV is contoured.

Use of image guided intensity modulated radiotherapy (IG-IMRT) preferably with rotational IMRT is mandatory. 3D image guidance (Cone Beam CT (CBCT) or equivalent image guidance) before each EBRT fraction is mandatory. This allows for use of reduced PTV margins (5mm from ITV45). The dose to the PTV45 should be homogenous, with at least 95% of the PTV covered by the 95% prescription isodose, and dose maximum less than 107% of the prescribed dose. Special attention is needed for the OAR irradiation in close proximity to the CTV-T HR (bladder, rectum, sigmoid and bowel). A help contour with a margin of 10 mm is generated around the CTV-T HR (CTV-T HR +10mm). The dose within this help contour should be less than 103% of 45Gy to avoid hotspots in OAR walls which are likely to also receive considerable BT dose. Lymph nodes will be boosted by simultaneous integrated boost (SIB) technique. Use of coverage probability (CoP) dose planning principles for lymph node boosting is mandatory.

Although institutional practise for nodal boosting and dose levels can be followed, the recommendation given within this protocol for the nodal boost is that total EBRT + BT dose should preferably be in the range 55-60 Gy EQD2.Total dose to PTV-Ns of about 60 Gy EQD2 can be achieved with the following fractionation schedules:

* Inside true pelvis: EBRT with SIB 25x2.2Gy= 55Gy physical dose. This schedule is equivalent to 56 Gy EQD2 EBRT + 3-4 Gy EQD2 from BT which results in a total dose of ~60 Gy EQD2.
* Outside true pelvis: EBRT with SIB 25x2.3Gy =57.5 Gy physical dose. This schedule is equivalent to ~59 Gy EQD2 and BT dose contribution is negligible.

All patients should receive concurrent weekly cisplatin (40 mg/m2) during the 5 weeks of EBRT, based on standard institutional protocol. If possible, it may be advantageous to initiate EBRT and concomitant chemotherapy in the beginning of a week to avoid loss of 2 days in overall treatment time (OTT) already during the first weekend.

EBRT is followed by MRI guided adaptive brachytherapy (IGABT). The overall treatment time (OTT), defined from the first external beam fraction to the final external beam or brachytherapy fraction dose is delivered should be < 50 days. To obtain maximal regression the treatment should always be initiated with EBRT and concomitant chemotherapy for 4-5 weeks before BT is applied in weeks. Systematic use of combined intracavitary and interstitial applicators (based on individual mould, ring, ovoids) is a preferred approach for appropriate dose adaptation which is dose escalation in particular for advanced parametrial disease and/or dose sparing in adjacent organs at risk. The first BT fraction has to be planned based on MRI with applicator in situ. Contouring for both tumour and OAR is performed for each insertion/implant of BT applicators by contouring on T2 weighted (para)-transversal MRI sequences in a dedicated 3D brachytherapy dose-planning system according to the GEC ESTRO Recommendations and the ICRU-89 report. Soft and hard dose planning constraints are detailed in the protocol. Doses are expressed as total EBRT and BT dose (each converted to EQD2). Hard constraints should be achieved in at least 90-95% of patients (per parameter), whereas soft constraints should be achieved in at least 70-80% of patients (per parameter). The priorities and balance between different DVH parameters are based on the therapeutic priorities (chance of tumor control versus risk of morbidity) as well as the level of evidence of dose effect for a given endpoint. Dose recording and reporting follows the recommendations of ICRU-89 report.

Standard of care CRT will be combined with the following study drugs:

Pembrolizumab: 5 intravenous administrations of Pembrolizumab (200 mg) every 3 weeks with the first administration at the start of chemoradiotherapy, followed by subsequent doses of 400 mg IV Pembrolizumab at 6 weeks intervals, starting week 16 up to week 102 with a maximum of 15 cycles. Pembrolizumab may be withheld after 1st year (week 54) in case of no evidence of disease. Lenvatinib: the combination with Lenvatinib will start after recovery of CRT, along with the 6 weekly cycles of Pembrolizumab, e.g. around 8-9 weeks after brachytherapy (week 16), at a dose of 20 mg daily oral and will continue up to week 48. Patients will be provided with a dosing card for Lenvatinib to complete during the treatment period. All patients will be asked to fill the dosing card once daily at the time of administrating Lenvatinib. It will include following information: dosing date, dose, dosing time, dosing missed and reason of missed dosing. They will be asked to bring the dosing card, along with their used medication packs, during their subsequent visit and will be used to assess compliance.

Haematology parameters and organ function will be checked through blood tests prior to each administration of Pembrolizumab and urine analysis prior to every other administration.

Tumor imaging is preferred to be acquired by computed tomography (CT) for uniform response evaluation. For the abdomen and pelvis, contrast-enhanced magnetic resonance imaging (MRI) may also be used when CT with iodinated contrast is contraindicated, or when local practice mandates it. MRI is the preferred modality for imaging the primary tumor when indicated. Initial tumor imaging at pre-screening (MRI and CT) must have been performed within 28 days prior to the date of registration. The site study team must review pre-treatment images to confirm the participant has measurable disease per RECIST 1.1 at diagnosis. Tumor imaging performed as part of routine clinical management is acceptable for use as screening tumor imaging if they are of diagnostic quality and performed within 28 days prior to the date of registration. Follow-up tumor imaging should be performed as per standard clinical practice. MRI is performed at 3 months and at 12 months (SOC), CT thorax/abdomen is performed at 12, 24 and 36 months. Based on clinical indications MRI may be repeated at 6 months (SOC).

Ethical considerations Ethical considerations relating to the clinical trial including the expected benefit to the individual subject or group of patients represented by the trial subjects as well as the nature and extent of burden and risks Pembrolizumab and Lenvatinib are cancer drugs that have proven to be effective against other cancers, both alone and in combination, such as for uterine cancer. Pembrolizumab also works well in combination with chemotherapy for advanced or metastatic cervical cancer and has been shown to be beneficial during and after chemoradiation for locally advanced cervical cancer. The study hypothesizes that over and above concurrent and Pembrolizumab monotherapy, the addition of Lenvatinib administered after CRT and brachytherapy will lead to improved outcomes in this population of locally advanced cervical cancer patients that are deemed to be at high risk of recurrence based on established risk factors.

Pembrolizumab and Lenvatinib may cause side effects (detailed in the protocol). Patients may experience side effects that can sometimes be serious or life-threatening, and/or side effects that may occur after you stopping Pembrolizumab. The side effects can occur in several tissues and organs at the same time. The following side effects of Pembrolizumab are common (may affect more than 10-20 people in 100 people receiving Pembrolizumab): Itchy skin; loose or watery stools, diarrhea, cough. The following side effects with Lenvatinib are common (may affect more than 1 in 10 people): high blood pressure; bleeding; bladder irritation or discomfort (cystitis); weight loss; diarrhoea.

Apart from side effects of the study drugs, taking part in the study will cost patients extra time, requires more and potentially longer stays in the hospital, and involves some discomfort from the additional measurements that are part of the study.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* High risk defined by either of the criteria:

  1. Squamous cell carcinoma FIGO 2018 stage IIIA, IIIB, IIIC1-IIIC2 OR
  2. Adenocarcinoma or adeno-squamous carcinoma Stage IB3-IIIC2.
* Have adequate haematological parameters and organ function as defined in the protocol Table 3.
* Have adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mm Hg.
* Have measurable disease based on RECIST 1.1 on imaging at diagnosis.
* The participant provides written informed consent for the trial.
* Patients should have been planned for radical chemoradiation and MR guided adaptive brachytherapy with intended treatment completion within 50 days.
* Patients should be deemed suitable for start of Pembrolizumab during chemoradiation and brachytherapy, and for start of Lenvatinib/Pembrolizumab 8 weeks after last brachytherapy as per local investigators assessment.
* Criteria for known Hepatitis B and C positive subjects:

Hepatitis B and C screening tests are not required unless:

* Known history of HBV or HCV infection
* As mandated by local health authority

Hepatitis B positive subjects:

* Participants who are HBsAg positive are eligible if they have received HBV antiviral therapy for at least 4 weeks and have undetectable HBV viral load prior to inclusion.
* Participants should remain on anti-viral therapy throughout study intervention and follow local guidelines for HBV anti-viral therapy post completion of study intervention.
* Participants with history of HCV infection are eligible if HCV viral load is undetectable at screening.
* Participants must have completed curative anti-viral therapy at least 4 weeks prior to randomization.

Exclusion Criteria:

* Patients with locally advanced cervical cancer and signs of organ wall involvement on MRI or non-gastrointestinal fistula.
* Major surgery within 3 weeks prior to first dose of study interventions. Brachytherapy is not considered a major surgery.
* Urine protein ≥1 g/24 hours. Note: Participants with proteinuria ≥2+ (≥100 mg/dL) on urine dipstick testing (or urinalysis) will undergo 24-hour urine collection for quantitative assessment of proteinuria.
* If a MUGA or cardiac ultrasound was performed (on clinical indication): having a LVEF below the institutional (or local laboratory) normal range.
* Radiographic evidence of encasement or invasion of a major blood vessel, or of intratumoral cavitation NOTE: the degree of proximity to major blood vessels should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following Lenvatinib therapy.
* Prolongation of QTcF interval to >480 ms. NOTE: If the QTcF is prolonged to >480 ms in the presence of a pacemaker, contact the Sponsor to determine eligibility.
* Clinically significant cardiovascular disease within 12 months from first dose of study intervention, including New York Heart Association Class III or IV congestive heart failure, unstable angina, myocardial infarction, cerebral vascular accident, or cardiac arrhythmia associated with hemodynamic instability.

Note: Medically controlled arrhythmia would be permitted.

* Gastrointestinal malabsorption or any other condition that might affect the absorption of Lenvatinib.
* Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
* WOCBP who has a positive urine pregnancy test within 72 hours prior to adjuvant phase. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. Note eligible patients for this trial are not WOCBP due to treatment with CRT.
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Known additional malignancy that is progressing or has required active treatment within the past 3 years.

Note: Participants with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ, excluding carcinoma in situ of the bladder, that have undergone potentially curative therapy are not excluded.

* Severe hypersensitivity (≥Grade 3) to Pembrolizumab or Lenvatinib and/or any of its excipients.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment and is allowed.
* History of (non-infectious) pneumonitis/interstitial lung disease that required steroids or has current pneumonitis/interstitial lung disease.
* Active infection requiring systemic therapy.
* Known history of Human Immunodeficiency Virus (HIV) infection. Note: No HIV testing is required unless mandated by local health authority.
* Known concurrent active Hepatitis B (defined as HBsAg positive and detectable HBV DNA) and/or Hepatitis C virus (defined as anti-HCV Ab positive and detectable HCV RNA [qualitative]) infection. See inclusion criteria 10

Note: no testing for Hepatitis B and Hepatitis C screening tests are not required unless:

* Known history of HBV and HCV infection
* As mandated by local health authority.

  * Has a history or current evidence of any condition, therapy, or laboratory abnormality or other circumstance that might confound the results of the study, interfere with the participant's participation for the full duration of the study, or such that it is not in the best interest of the participant to participate, in the opinion of the treating investigator.
  * Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
  * Has had an allogenic tissue/solid organ transplant.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | From date of enrollment to 24 months
  Actuarial Progression free survival (PFS) rate at 24 months, with a PFS event defined by either progression, using investigator assessed RECIST 1.1, or by death from any cause.

SECONDARY OUTCOMES:
Overall Survival | From date of enrollment to 24 and to 36 months
  Actuarial Overall Survival (OS) rate at 24 and at 36 months, with an OS event defined as death by any cause.
Progression Free Survival | From date of enrollment to 36 months
  Actuarial Progression free survival (PFS) rate at 36 months, with a PFS event defined by either progression, using investigator assessed RECIST 1.1, or by death from any cause.
Local Control | From date of enrollment to 24 and to 36 months.
  Actuarial rate of Local Control (LC) of the primary tumor at 24 and 36 months, with an event defined as absence of tumor at the level of the cervix, detected at gynecological examination or imaging, and histological confirmed.
Regional Nodal Control | From date of enrollment to 24 and to 36 months.
  Actuarial rate of Regional Nodal Control at 24 and 36 months, with an event defined as absence of pathological pelvic and / or para-aortic lymph node involvement assessed by imaging.
Adverse Events | From date of enrollment to 24 and 36 months.
  Adverse Events defined and graded by CTCAE v 5.0, crude and actuarial rates at 24 and 36 months.
Patient reported symptoms and health related quality of life | At baseline prior to the start of treatment, at 5 weeks after start of treatment, at the first 6 weekly cycle of pembrolizumab, at 3, 6, 9, 12, 24, 36, 48 and 60 months.
  Patient reported symptoms and health related quality of life are determined using the validated EORTC QLQC30 and Cx-24 questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided